CLINICAL TRIAL: NCT04640818
Title: Safety and Efficacy of a Therapy With Cladribine Following a Treatment With Anti CD20 Compounds in Relapsing Multiple Sclerosis Patients: a Pilot Study
Brief Title: Safety and Efficacy of Cladribine Therapy After Anti CD20 Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Claudio Gobbi (Other Government)
Collaborators: Merck AG Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Claudio Gobbi, Head Physician, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Other Study IDs: EOCNSIMS.2001
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: anti CD20 therapy; cladribine
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine; Rituximab; ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CLAD-GROUP: Patients with cladribine therapy
  Interventions: Drug: Cladribine Oral Tablet
- CD20-GROUP: Patients with anti CD20 therapy (ocrelizumab or rituximab)
  Interventions: Drug: Rituximab; Drug: Ocrelizumab

INTERVENTIONS:
Drug: Cladribine Oral Tablet — Treatment according to the label and medical prescription
  Other Names: Mavenclade
  Groups: CLAD-GROUP
Drug: Rituximab — Treatment according to the label and medical prescription
  Other Names: Mabthera, Rixathon
  Groups: CD20-GROUP
Drug: Ocrelizumab — Treatment according to the label and medical prescription
  Other Names: Ocrevus
  Groups: CD20-GROUP

SUMMARY:
Prolonged anti CD20 therapy for the treatment of active multiple sclerosis leading to continuous B cell depletion is associated with hypogammaglobulinemia predisposing to a potentially increased risk of serious infections, particularly in the more disabled and aged patients. No data have been published on the sequential use of anti CD20 therapies and cladribine, that is thought to act as an immune reconstitution agent. his study aims at investigating IgG and IgM serum concentration changes at 6 and 12 months after switching to cladribine in patients previously treated with anti CD20 therapies (ie, ocrelizumab ≥1.8 gr or rituximab 3.0 gr) for ≥18 months, as compared to continued anti CD20 therapies.

DETAILED DESCRIPTION:
The study population will include patients with remitting relapsing multiple sclerosis consulting the Multiple Sclerosis Center of Neurocenter of Southern Switzerland.

Enrolled patients will have 5 Study Visits, one every 3 months according to clinical practice. At visits at 3 and 6 months only adverse events will be collected for study purposes. Clinical assessments will be performed at baseline, Month 6 and Month 12. Clinical assessments correspond to medical exams performed routinely in MS patients treated with anti CD20 or cladribine therapy: clinical assessments, monitoring haemoglobin parameters, serum immunoglobulins, liver and renal function.(6, 12 months), radiological disability progression and biomarker of ongoing neurodegeneration (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Relapsing MS according to Lublin;
* Treatment with ocrelizumab or rituximab for ≥18 months and having received 1.8 / 3.0 gr, respectively;
* CLAD_GROUP: Planning to switch to cladribine because of concerns about increased risks of infections related to hypogammaglobulinemia developing during long term anti CD20 therapies or a documented decrease of ≥10% IgG and/or IgM compared to pre- anti CD20 therapy;
* or CD20_GROUP: no need to stop CD20 therapy due decrease of ≥10% IgG and/or IgM, or increased risk of infections related to hypogammaglobulinemia or other reasons, continued anti CD20 therapies clinically indicated;
* EDSS ≤7.0;
* Age >18 years.

Exclusion Criteria:

* Non relapsing MS;
* Pregnancy - breastfeeding;
* Contraindications to perform MRI;
* Contraindication to receive cladribine or to continue anti CD therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in IgG serum concentrations in Cald-Group | 6 months
  Standard laboratory test
Changes in IgM serum concentrations in Cald-Group | 6 months
  Standard laboratory test
Changes in IgG serum concentrations in Clad-Group | 12 months
  Standard laboratory test
Changes in IgM serum concentrations in Clad-Group | 12 months
  Standard laboratory test

SECONDARY OUTCOMES:
Changes in IgG serum concentrations after switching to cladribine, as compared to continued anti CD20 therapies | 6 months
  Standard laboratory test
Changes in IgM serum concentrations after switching to cladribine, as compared to continued anti CD20 therapies | 6 months
  Standard laboratory test
Changes in IgG serum concentrations after switching to cladribine, as compared to continued anti CD20 therapies | 12 months
  Standard laboratory test
Changes in IgM serum concentrations after switching to cladribine, as compared to continued anti CD20 therapies | 12 months
  Standard laboratory test
Proportion of patients reaching NEDA -3 | 12 months
  NEDA -3: no relapses, no disability progression, no new/enlarging or Gd enhancing brain or spinal MR lesions
Annualized relapse rate (ARR) over 12 months after switching to cladribine as compared to patients continuing anti CD20 therapies | 12 months
  ARR will be calculated based on recorded number of relapses
Proportion of patients with disability progression | 6 months
  Expanded disability scale 0-6 (6 worst outcome)
Proportion of patients with disability progression | 12 months
  Expanded disability scale 0-6 (6 worst outcome)
Number/volume of cumulative new T2/ enlarging lesions at brain and spinal MRI over 12 months after switching to cladribine, as compared to patients continuing anti CD20 therapies | 12 months
  Evaluation of MRI
Number/volume of cumulative Gd enhancing lesions at brain and spinal MRI over 12 months after switching to cladribine, as compared to patients continuing anti CD20 therapies | 12 months
  Evaluation of MRI
Changes in serum neurofilament light chain concentration | 12 months
  single-molecule array (Simoa) assay

OTHER OUTCOMES:
Frequency of infections | 6 months
  Safety endpoint
Frequency of infections | 12 months
  Safety endpoint
Intensity of infections | 6 months
  Safety endpoint, intensity will be rated according to the following definitions:
  Mild: Awareness of a sign or symptom that does not interfere with the study participant's usual activity or is transient, resolved without treatment and with no sequelae; Moderate: Interferes with the study participant's usual activity and/or requires symptomatic treatment; Severe: Symptom(s) causing severe discomfort and significant impact of the study participant's usual activity and requires treatment.
  Serious: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, or is otherwise considered as medically important.
Intensity of infections | 12 months
  Safety endpoint, intensity will be rated according to the following definitions:
  Mild: Awareness of a sign or symptom that does not interfere with the study participant's usual activity or is transient, resolved without treatment and with no sequelae; Moderate: Interferes with the study participant's usual activity and/or requires symptomatic treatment; Severe: Symptom(s) causing severe discomfort and significant impact of the study participant's usual activity and requires treatment.
  Serious: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, or is otherwise considered as medically important.
Proportion of patients with abnormal creatinine values of clinical relevance | 6 months
  Safety endpoint
Proportion of patients with abnormal creatinine values of clinical relevance | 12 months
  Safety endpoint
Proportion of patients with abnormal ASAT values of clinical relevance | 6 months
  Safety endpoint
Proportion of patients with abnormal ASAT values of clinical relevance | 12 months
  Safety endpoint
Proportion of patients with abnormal ALAT values of clinical relevance | 6 months
  Safety endpoint
Proportion of patients with abnormal ALAT values of clinical relevance | 12 months
  Safety endpoint
Proportion of patients with any abnormal hematology values of clinical relevance | 6 months
  Safety endpoint
Proportion of patients with any abnormal hematology values of clinical relevance | 12 months
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gobbi, MD, Principal Investigator — Ospedale Regionale di Lugano, Neurocentro della Svizzera italiana, Centro Sclerosi multipla
Locations (1):
- Neurocenter of Southern Switzerland, Ospedale Regionale di Lugano, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No